CLINICAL TRIAL: NCT07334262
Title: A Study to Evaluate the Food Effect on the Pharmacokinetics of RNK08954 Tablets and to Assess the Mass Balance of [14C]RNK08954 in Healthy Adult Male Subjects in China
Brief Title: A Study to Evaluate the Food Effect on RNK08954 in Healthy Participants, and the Mass Balance Study of [14C]RNK08954 in Healthy Adult Male Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ranok Therapeutics (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ranok Therapuetics Co. Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RNK08954-03
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Food Effect; Mass Balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNK08954 Treatment A (Experimental): 1200mg RNK08954, following an overnight fast of at least 10 hours
  Interventions: Drug: RNK08954
- RNK08954 Treatment B (Experimental): 1200mg RNK08954, administered 30 minutes after the start of a high-fat/high-calorie meal breakfast.
  Interventions: Drug: RNK08954

INTERVENTIONS:
Drug: RNK08954 — KRAS G12D inhibitor

SUMMARY:
An Study of Orally Administered RNK08954 in Healthy Adult Subjects to Determine the Effect of Food on the Pharmacokinetics of RNK08954，Mass Balance Study of [14C] RNK08954 in Chinese Healthy Adult Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18-45 years of age, inclusive, at the screening visit.
* Male participants must have a body weight of no less than 50 kg, and female participants must have a body weight of no less than 45 kg. The Body mass index (BMI) should be between 19 and 26 kg/m² (inclusive).
* Must follow protocol specified contraception guidance.
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

* Clinically significant abnormalities found in comprehensive physical examinations, vital signs, laboratory tests, 12-lead electrocardiogram, chest X-ray, etc.
* Positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or treponema pallidum antibody.
* Individuals with allergic constitution.
* Any history of clinically significant diseases or conditions that, in the investigator's judgment, may affect the trial results.
* History or family history of organic heart disease, heart failure, myocardial infarction, angina pectoris, torsades de pointes, ventricular tachycardia, QT prolongation syndrome.
* Gastrointestinal diseases that cause clinically significant symptoms such as nausea, vomiting, diarrhea, or malabsorption syndrome, or those with a history of vomiting or diarrhea within one week prior to screening.
* Individuals with dysphagia.
* Undergone major surgery within six months prior to the first dose or whose surgical incision has not fully healed.
* Used investigational drugs or received other experimental treatments within three months prior to the first dose or are currently participating in any other interventional clinical trials.
* Vaccinated within one month prior to the first dose or plan to be vaccinated during the trial period.
* Used any drugs affecting drug-metabolizing enzymes or transporters within 30 days prior to the first dose.
* Taken any prescription drugs, over-the-counter medications, herbal medicines, or dietary supplements within 14 days prior to the first dose.
* Smoke more than 10 cigarettes per day or habitually use nicotine-containing products within three months prior to the first dose.
* Current or previous alcohol abuse, or frequent alcohol consumption within six months prior to the first dose, or those with a positive alcohol breath test.
* History of drug abuse, use of soft drugs within three months prior to the first dose, or use of hard drugs within one year prior to the first dose, or those with a positive urine drug abuse screening.
* Individuals who habitually or excessively consume grapefruit juice, tea, coffee, and/or caffeinated beverages.
* History of blood loss or blood donation (≥400 mL) within three months prior to the first dose, those who have received blood transfusions or blood products within one month prior to the first dose, or those who plan to donate blood within three months after the trial.
* Special dietary requirements, intolerance to high-fat meals, or inability to comply with a standardized diet.
* History of needle or blood phobia, difficulty with blood collection, or intolerance to venipuncture.
* Pregnant or lactating women.
* have poor compliance or other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Plasma Pharmacokinetics (PK) of a single dose of RNK08954 after a standardized high-fat/high-calorie meal and after fasting: Tmax | 30 days
  Time of Maximum concentration (Tmax)
Plasma Pharmacokinetics (PK) of a single dose of RNK08954 after a standardized high-fat/high-calorie meal and after fasting: Tlag | 30 days
  absorption lag-time (Tlag)
Plasma Pharmacokinetics (PK) of a single dose of RNK08954 after a standardized high-fat/high-calorie meal and after fasting: Cmax | 30 days
  Cmax for RNK08954 administered with and without food.
Plasma Pharmacokinetics (PK) of a single dose of RNK08954 after a standardized high-fat/high-calorie meal and after fasting: AUC0-inf | 30 days
  Area under plasma Concentration (AUC) from zero to infinity
Plasma Pharmacokinetics (PK) of a single dose of RNK08954 after a standardized high-fat/high-calorie meal and after fasting: AUC0-last | 30 days
  Area Under the concentration-time Curve from time zero to the time of the last

SECONDARY OUTCOMES:
Incidence,frequency and severity of adverse events (AEs）of RNK08954 as assessed by CTCAE 5.0 | 30 days
  As a measure of the safety and tolerability of RNK08954 the number of subjects who experienced any treatment emergent AE (TEAE), any causally related AE, any serious AE (SAE), and any causally related SAE are presented.
Electrocardiogram (ECG) parameters: HR, PR, QRS, QT, and QTc | 30 days
  Safety and tolerability measures will be recorded at the indicated timepoints
Systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHG) | 30 days
  Safety and tolerability measures will be recorded at the indicated timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China